CLINICAL TRIAL: NCT05917379
Title: The Safety and Efficacy of Fecal Microbiota Transplantation in Patients With Chronic Insomnia Disorder
Brief Title: The Efficacy and Safty of FMT in Patients With CID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Gao Teng, Peking University, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUSH 20241218
Record Dates: First submitted 2023-05-25; First posted 2023-06-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Insomnia Chronic; Fecal Microbiota Transplantation; Sleep Disorder; Depression; Anxiety; Cognitive Impairment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Depression; Anxiety Disorders; Cognitive Dysfunction | interventions — Fecal Microbiota Transplantation; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Experimental): Investigators have 2 subgroups here, pure Fecal microbiota transplantation-F: Fecal microbiota capsules(0.75g stool/capsule) (60 capsules), within 3 days, another 20 fecal microbiota capsules(0.75g stool/capsule) at week 2. Additionally, they will take placebo B for 45 days from the beginning; Fecal microbiota transplantation+synbiotics-M: Fecal microbiota capsules(0.75g stool/capsule) (60 capsules), within 3 days, another 20 fecal microbiota capsules(0.75g stool/capsule) at week 2. Additionally, they will take synbiotics (Lactobacillus Helveticus Bifidobacterium longum + inulin) (3g/day) for 45 days from the beginning.
  Interventions: Biological: fecal microbiota; Dietary Supplement: synbiotics
- Non-FMT (Placebo Comparator): Investigators have 2 subgroups here, synbiotics control-S: PlaceboA capsules (60 capsules), within 3 days, another 20 placeboA capsules(0.75g stool/capsule) at week 2. Additionally, they will take synbiotics (Lactobacillus Helveticas+ Bifidobacterial longum + inulin) (3g/day) for 45 days from the beginning; Double Placebo-P: PlaceboA capsules (60 capsules), within 3 days, another 20 placeboA capsules(0.75g stool/capsule) at week 2. Additionally, they will take placebo B for 45 days from the beginning.
  Interventions: Other: Placebo; Dietary Supplement: synbiotics

INTERVENTIONS:
Biological: fecal microbiota — FMT utilizes stool from a healthy donor and puts them into capsules after processing
  Other Names: FMT
  Arms: FMT
Other: Placebo — Starch into the same outlook capsule with fecal microbiota
  Arms: Non-FMT
Dietary Supplement: synbiotics — Lactobacillus Helveticas+ Bifidobacterial longum + inulin(3g/day)

SUMMARY:
This clinical trial aims to learn about the efficacy of fecal microbiota transplantation in patients with chronic insomnia disorder. The main question[s] it aims to answer is:

• Effectiveness of the FMT oral capsule route for patients with chronic insomnia Participants in the intervention group will be given FMT by boral capsule pathway, and in the control group, they will be given the same appearance capsules containing starch.

Researchers will compare the sleep status(PSQI and PSG)of the patients in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed CID by DSM-5
2. 18-60 years old24
3. Body Mass Index (BMI) within the range of 18-24 kg/m²
4. No other pharmacologic treatment in the last month or at the stable maintenance stage (stable dose for more than two months)

Exclusion Criteria:

1. Currently pregnant, planning pregnancy shortly, or breastfeeding
2. Undergoing or recently received immunosuppressive therapy, or severe immunosuppression (neutrophil count <1500 cells/mm³, lymphocyte count <500 cells/mm³)
3. Diagnosis of one or more specific gastrointestinal disorders (e.g., Crohn's disease, ulcerative colitis, gastrointestinal tumors, pseudomembranous enteritis, gastrointestinal bleeding, enterocutaneous fistula, etc.)
4. Diseases with significant correlations to gut microbiota include Type 2 Diabetes, thyroid disorders, migraines, and autoimmune diseases
5. Ex-/intraintestinal organ infection
6. Abnormal liver or kidney function
7. Faecal occult blood test (+)
8. Suffering from chronic pain, restless leg syndrome, obstructive sleep apnea, or thyroid disorders.
9. Central nervous system disorders (e.g., epilepsy, Parkinson's disease, history of traumatic brain injury, cerebrovascular diseases, etc.)
10. Current smokers or alcohol drinkers
11. History of food or antibiotic allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | 1 month post FMT
  (Total Time Asleep / Total Time in Bed×100%) of CID patients will be objectively ，assessed using PSG at week 4 post-FMT (compared to baseline). Additionally, subjective measures including PSQI and ISI scores will be included

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index，PSQI | baseline and 1-, 2-, 3-, 6- months post FMT
  The PSQI was used to assess the sleep quality of the participants in the last 1 month. It consists of 19 self-assessments and 5 self-assessment items, of which the 19th self-assessment item and 5 self-assessment items do not participate in the scoring. The 18 items formed 7 components, and each component was scored according to 0-3 levels. The cumulative score of PSQI total score ranged from 0 to 2 l. The higher the score, the worse the sleep quality
Insomnia Severity Index，ISI | baseline and 1-, 2-, 3-, 6- months post FMT
  ISI is a commonly used insomnia severity scale used to assess the extent and impact of individual insomnia in the past two weeks. The ISI consists of seven items, and individuals need to choose the answer best suitable for their condition on each item, and then aggregate the scores of all items to get the total score. The total score ranged from 0 to 28, with higher scores indicating higher insomnia severity. Each item has four answer options, used to describe the frequency of insomnia, severity and effects on the individual.
Bray-Curtis dissimilarity | baseline and 1-month post FMT
  Bray-Curtis dissimilarity is a beta diversity metric used to quantify differences in microbial community composition between two time points. A higher dissimilarity score indicates greater divergence in taxonomic profiles. This outcome measures the change in gut microbiota structure from baseline to 1-month after fecal microbiota transplantation (FMT), serving as an index of engraftment and microbial shift
Sleep onset latency (SL) | baseline and 1 month post FMT
  Based on polysomnography (mins)
Self-Rating Anxiety Scale (SAS) | baseline and 1-, 2-, 3-, 6- months post FMT
  Participants need to according to the past a period of time (usually in the past week or two weeks), choose a most accord with their feelings answer options, usually expressed by the following level: no or little time (1), part of the time (2 points), quite a large amount of time (3 points), most or all of the time (4 points). An initial assessment of individual anxiety was possible by calculating the total score.
Self-Rating Depression Scale (SDS) | baseline and 1-, 2-, 3-, 6-months post FMT
  It usually contains 20 topics and is widely used in research and clinical practice. Participants need to according to the past a period of time (usually in the past week or two weeks), choose a most accord with their feelings answer options, usually expressed by the following level: no or little time (1), part of the time (2), quite a large amount of time (3), most or all of the time (4). The total raw score ranges from 20 to 80, and is typically converted to a standard score by multiplying by 1.25 (range: 25 to 100), with higher scores indicating greater severity of depression.
Gastrointestinal Symptom Rating Scale，GSRS | baseline and 1-, 2-, 3-, 6-months post FMT
  The GSRS includes 15 questions about gastrointestinal symptoms covering a range of symptoms including abdominal pain, flatulence, nausea, vomiting, loss of appetite, etc.The score rang from 16-112, the less the better.
Arousal index (ArI) | baseline and 1-month post FMT
  Based on polysomnography (events/h)
Non-rapid eye movement sleep duration(NREM) | baseline and 1-month post FMT
  Based on polysomnography (mins)
Rapid eye movement sleep duration(REM) | baseline and 1-month post FMT
  Based on polysomnography (mins)
Observed OTUs | baseline and 1-month post FMT
  Observed OTUs (Operational Taxonomic Units) represent the count of unique taxa identified in a sample, reflecting species richness. This outcome measures the number of observed OTUs in fecal samples at baseline and 1-month post-FMT, indicating changes in microbial richness following intervention.
Shannon Diversity Index | baseline and 1-month post FMT
  The Shannon index is a commonly used α-diversity metric that accounts for both richness and evenness in microbial communities. Higher values reflect greater diversity. This outcome evaluates within-sample microbial diversity before and after FMT.
Simpson Diversity Index | baseline and 1-month post FMT
  The Simpson index measures the probability that two randomly selected individuals in a sample belong to the same species. It is sensitive to dominant taxa. This outcome assesses within-sample microbial diversity changes induced by FMT.
Chao1 Richness Estimator | baseline and 1-month post FMT
  The Chao1 index estimates microbial species richness by accounting for the number of rare taxa (singletons and doubletons). It provides a more robust estimate of total richness compared to observed OTUs. This outcome evaluates the estimated richness change after FMT.

OTHER OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status，RBANS | baseline and 3-month post FMT
  The RBANS consists of 12 subtests that assess five cognitive domains: immediate memory, visuospatial/constructional ability, language, attention, and delayed memory. It yields a Total Scale Index Score with a mean of 100 and a standard deviation of 15, where higher scores indicate better cognitive performance.
  RBANS is widely used in clinical and research settings to evaluate cognitive impairment, monitor disease progression, and assess treatment effects. Individual scores can be compared with normative data stratified by age and education level.
Heart Rate Variability ,HRV | baseline and 1 months post FMT
  Heart rate variability is where the amount of time between your heartbeats fluctuates slightly. Even though these fluctuations are undetectable except with specialized devices, they can still indicate current or future health problems, including heart conditions and mental health issues like anxiety and depression.
Multiplex cytokine analysis(pg/mL) | baseline and 1-month post FMT
  IL-1β, IL-6
Ach levels（pmol/mL） | baseline and 1-month post FMT
  Automatic nervous system related factors
NE levels（pg/mL） | baseline and 1-month post FMT
  Automatic nervous system related factors

CONTACTS AND LOCATIONS:
Overall Officials: Lu, Study Director — Peking University six hospital
Locations (1):
- Peking University Six Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the research results, the data will be shared on this website and relevant journal platforms
Supporting Information: Study Protocol
Time Frame: 1st December 2025
Access Criteria: Open assess

REFERENCES:
- [Background] Wang Z, Wang Z, Lu T, Chen W, Yan W, Yuan K, Shi L, Liu X, Zhou X, Shi J, Vitiello MV, Han Y, Lu L. The microbiota-gut-brain axis in sleep disorders. Sleep Med Rev. 2022 Oct;65:101691. doi: 10.1016/j.smrv.2022.101691. Epub 2022 Aug 31. PMID 36099873
- [Background] Wang X, Wang Z, Cao J, Dong Y, Chen Y. Gut microbiota-derived metabolites mediate the neuroprotective effect of melatonin in cognitive impairment induced by sleep deprivation. Microbiome. 2023 Jan 31;11(1):17. doi: 10.1186/s40168-022-01452-3. PMID 36721179
- [Background] Perlis ML, Posner D, Riemann D, Bastien CH, Teel J, Thase M. Insomnia. Lancet. 2022 Sep 24;400(10357):1047-1060. doi: 10.1016/S0140-6736(22)00879-0. Epub 2022 Sep 14. PMID 36115372
- [Background] Li Y, Zhang B, Zhou Y, Wang D, Liu X, Li L, Wang T, Zhang Y, Jiang M, Tang H, Amsel LV, Fan F, Hoven CW. Gut Microbiota Changes and Their Relationship with Inflammation in Patients with Acute and Chronic Insomnia. Nat Sci Sleep. 2020 Nov 5;12:895-905. doi: 10.2147/NSS.S271927. eCollection 2020. PMID 33177907
- [Background] Haifer C, Kelly CR, Paramsothy S, Andresen D, Papanicolas LE, McKew GL, Borody TJ, Kamm M, Costello SP, Andrews JM, Begun J, Chan HT, Connor S, Ghaly S, Johnson PD, Lemberg DA, Paramsothy R, Redmond A, Sheorey H, van der Poorten D, Leong RW. Australian consensus statements for the regulation, production and use of faecal microbiota transplantation in clinical practice. Gut. 2020 May;69(5):801-810. doi: 10.1136/gutjnl-2019-320260. Epub 2020 Feb 11. PMID 32047093
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878